CLINICAL TRIAL: NCT05673083
Title: Impact of a Health Technology Intervention on Patient Activation in Multiple Myeloma
Status: Active, not recruiting | Type: Observational
Sponsor: All4Cure (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: All4Cure02
Record Dates: First submitted 2022-12-22; First posted 2023-01-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma; Multiple Myeloma, Refractory; Multiple Myeloma With Failed Remission
Keywords: Multiple Myeloma; All4Cure; Patient Activation; PAM-13
MeSH Terms: conditions — Multiple Myeloma; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this pilot study is to evaluate the impact of All4Cure enrollment on patients with multiple myeloma. The main question it aims to answer are:

• Does All4Cure effect patient activation as assessed by the PAM-13 survey?

Participants will be asked to:

* fill out quarterly PAM-13 surveys through the All4Cure website to assess patient activation.
* fill out monthly Patient Reported Outcome (PRO) surveys through the All4Cure website.
* fill out a baseline and exit All4Cure surveys through the All4Cure website to assess patient perceptions of All4Cure at the beginning and the end of the study.

DETAILED DESCRIPTION:
The goal of this pilot study is to evaluate the impact of All4Cure enrollment on patients with multiple myeloma.

This study uses surveys to assess attitudes and perceptions of patients with myeloma at baseline and following their enrollment into All4Cure. The PAM-13 surveys will be administered at baseline and at 3-month intervals for a total of 5 surveys over 12 months. Patient attitudes and perceptions about the All4Cure platform will be assessed at baseline and at 12 months. Physicians caring for patients enrolled in this study will be surveyed twice -- at baseline and when all their patients have completed the study. Additionally, all patients will receive monthly surveys to assess symptoms associated with myeloma and its treatment using 36 survey items obtained from Patient Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE).

The study has the following objectives:

Primary objective To evaluate the impact of All4Cure enrollment on patients with multiple myeloma. The primary endpoint is the effect of All4Cure on patient activation, as assessed by the PAM-13 survey (change in results from baseline survey to the last completed survey).

Secondary objectives:

To evaluate the feasibility (i.e., ≥50% approach-to-enrollment rate of eligible participants and ≥70% completion of at least two PAM-13 surveys over a 12-month period) and acceptability (i.e., ≤20% withdrawing from the study and ≤20% withdrawing from All4Cure) of participation in All4Cure's digital platform for survivors with multiple myeloma.

To evaluate associations between participant activation levels (as assessed by PAM-13) and symptom burden, as measured by the Patient Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE).

To evaluate patient expectations and perceptions of the utility of All4Cure in their care and their association with PAM-13 results.

To evaluate associations between patient participation in the All4Cure platform (e.g. patient visits to the platform, patient posts on the platform, All4Cure posts on patient dashboards, and provision of MyelomaMap™ reports) and PAM-13 results.

To evaluate physician expectations and perceptions of the utility of All4Cure in their care of patients with multiple myeloma and their association with the PAM-13 results of their patients.

ELIGIBILITY:
Inclusion Criteria:

1. have a diagnosis of multiple myeloma.
2. are aged 18 years and older.
3. can read and e-consent to participate in the study.
4. can speak English.
5. can complete surveys at pre-specified intervals.
6. have access to a device that would allow for the completion of surveys (including at home, at work, at the oncologist's office or elsewhere).
7. are cared for by a physician who is enrolled in All4Cure.

Exclusion Criteria:

1. Patients will be excluded who are unable to engage with All4Cure or are already participants in All4Cure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll up to 200 patients with a diagnosis of multiple myeloma who are receiving treatment at Cancer Specialists of North Florida (CSNF, Florida), Northwest Medical Specialties (NWMS, Washington state), or Highlands Oncology Group (HOG, Arkansas).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patient Activation | 24 months
  Patient activation emphasizes patients' willingness and ability to take independent actions to manage their health and care. A widely used definition equates patient activation with understanding one's role in the care process and having the knowledge, skill, and confidence to manage one's health and health care. A growing body of evidence shows that patients who are more activated have better health outcomes and care experiences. This will be assessed through the PAM-13 survey which has a scale of 1-4, with 4 being the highest level of patient activation and associated with the best patient outcomes and 1 being the lowest level of patient activation.

SECONDARY OUTCOMES:
Evaluate associations between Patient Activation and symptom burden | 24 months
  Evaluate associations between participant activation levels (as assessed by PAM-13) and symptom burden, as measured by the Patient Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE).
Evaluate the feasibility and acceptability of participation in All4Cure's digital platform for survivors with multiple myeloma | 24 months
  evaluate the feasibility (i.e., ≥50% approach-to-enrollment rate of eligible participants and ≥70% completion of at least two PAM-13 surveys over a 12-month period) and acceptability (i.e., ≤20% withdrawing from the study and ≤20% withdrawing from All4Cure) of participation in All4Cure's digital platform for survivors with multiple myeloma.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Misson Cancer + Blood, Des Moines, Iowa
  - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oncology Consultants, Houston, Texas
  - Northwest Medical Specialties PLLC, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No